CLINICAL TRIAL: NCT01033890
Title: Local Anesthesia With Sedation for Cochlear Implant Surgery: 3 Case Report
Brief Title: Local Anesthesia With Sedation for Cochlear Implant Surgery
Acronym: IC
Status: Completed | Type: Observational
Sponsor: Instituto Paranaense de Otorrinolaringologia (Other)
Responsible Party: Principal Investigator, Rogerio Hamerschmidt, Professor, Instituto Paranaense de Otorrinolaringologia
Other Study IDs: IC-026; IPO IC 026 (Registry Identifier: IPO - IC 026); IPO - IC026
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cochlear Implant Surgery
Keywords: local anesthesia; cochlear implant; sedation; 3 patients submitted to cochlear implant surgery with local anesthesia with sedation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
ABSTRACT

Objectives: The aim of this article is to illustrate the possibility of performing a cochlear implant with local anesthesia and sedation, the anesthesic technique and the advantages of that in comparison to a general anesthesia.

Materials and method: The investigators describe two successful surgeries done with local anesthesia, including the neural telemetry and the conditions the patient presented after the surgery, with a very good recovery and no complications during and after the procedure.

Key words: local anesthesia, cochlear implant

ELIGIBILITY:
Inclusion Criteria:

* adult patients with total deafness

Exclusion Criteria:

* children under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 adult patients with total deafness
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Good liability and pos operative period of the patients submitted to cochlear implant surgery with local anestesia and sedation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Hamerschmidt, Principal Investigator — Instituto Paranaense de Otorrinolaringologia
Locations (1):
- Instituto Paranaense de Otorrinolaringologia, Curitiba, Paraná, Brazil